CLINICAL TRIAL: NCT02639611
Title: Effectiveness of Acupuncture in Post-Mastectomy Patients With Tissue Expanders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03266
Record Dates: First submitted 2015-12-22; First posted 2015-12-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast Expanders
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Post Operative Acupuncture Treatment (Active Comparator)
  Interventions: Other: Immediate Post Operative Acupuncture Treatment
- Acupuncture Treatment After 6 Weeks of Recovery (Active Comparator)
  Interventions: Other: No Acupuncture Treatment

INTERVENTIONS:
Other: Immediate Post Operative Acupuncture Treatment — acupuncture treatment immediately after surgery (twice a week for 6 weeks)
  Arms: Immediate Post Operative Acupuncture Treatment
Other: No Acupuncture Treatment — no acupuncture treatment for 6 weeks, but offered acupuncture at the end of the 6 week study period.
  Arms: Acupuncture Treatment After 6 Weeks of Recovery

SUMMARY:
The primary purpose of this study is to evaluate changes in shoulder tightness, chest tightness, and general pain related to post-mastectomy reconstructive surgery with tissue expansion in women who are randomized to receive acupuncture treatment immediately after surgery (twice a week for 6 weeks) compared to those who are randomized to no acupuncture treatment for 6 weeks, but offered acupuncture at the end of the 6 week study period.

ELIGIBILITY:
Inclusion Criteria:

* Women who are newly diagnosed with breast cancer, enrolled in the The Breast Cancer Database of NYU Cancer Center (BCD) and who are having breast cancer surgery involving a mastectomy procedure with insertion of a tissue expander for reconstructive purposes
* Women who are newly diagnosed with breast cancer
* Women who are enrolled in the Breast Cancer Database (BCD)
* Women who are having breast cancer surgery involving a mastectomy procedure with insertion of a tissue expander for reconstructive purposes

Exclusion Criteria:

* Women who had neoadjuvant chemotherapy and/or radiation therapy, women who are currently on anticoagulant therapy, women who are having breast reconstruction with Alloderm, women who have chronic pre-operative pain, and/or women who have had a history of previous implants or prior augmentations
* Women who had neoadjuvant chemotherapy and/or radiation therapy
* Women who are currently on anticoagulant therapy
* Women who are having breast reconstruction with Alloderm
* Women who have chronic pre-operative pain
* Women who have had a history of previous implants or prior augmentations
* Women who are currently on anticoagulant therapy
* Women who are having breast reconstruction with Alloderm
* Women who have chronic pre-operative pain
* Women who have had a history of previous implants or prior augmentations

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Shoulder Tightness Score on Pain and Discomfort Assessment Questionnaire | 6 Weeks
Chest Tightness Score on Pain and Discomfort Assessment Questionnaire | 6 Weeks
General Pain Score on Pain and Discomfort Assessment Questionnaire | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Freya Schnabel, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States